CLINICAL TRIAL: NCT02342795
Title: Randomized Controlled Trial Methods for Novel Tobacco Products Evaluation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Penn State University (Other); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HM20002759; 5P50DA036105-02 (NIH)
Record Dates: First submitted 2014-12-16; First posted 2015-01-21 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Nontherapeutic
MeSH Terms: interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- cigarette substitute (Experimental): The QuitSmart cigarette substitute is a plastic tube that looks like a real cigarette and is designed to provide the same draw resistance as a smoker's usual cigarette. There is no drug delivery with this product. Two cigarette substitutes and a product manual are provided to participants following randomization and replacement products are provided throughout the intervention period (24 weeks).
  Interventions: Other: cigarette substitute
- e-cigarette (with 0 mg/ml nicotine) (Experimental): The e-cigarette used will be the EGO e-cigarette (marketed by www.liquidexpress.com). Each participant randomized to an ECIG condition will receive 2 e-cigarette batteries, 1 wall adapter, 1 USB charger, and a user manual. Cartomizers containing 0 mg/ml nicotine will be provided throughout the intervention period (24 weeks).
  Interventions: Other: e-cigarette
- e-cigarette (with 8 mg/ml nicotine) (Experimental): The e-cigarette used will be the EGO e-cigarette (marketed by www.liquidexpress.com). Each participant randomized to an ECIG condition will receive 2 e-cigarette batteries, 1 wall adapter, 1 USB charger, and a user manual. Cartomizers containing 8 mg/ml nicotine will be provided throughout the intervention period (24 weeks).
  Interventions: Other: e-cigarette
- e-cigarette (with 36 mg/ml nicotine) (Experimental): The e-cigarette used will be the EGO e-cigarette (marketed by www.liquidexpress.com). Each participant randomized to an ECIG condition will receive 2 e-cigarette batteries, 1 wall adapter, 1 USB charger, and a user manual. Cartomizers containing 36 mg/ml nicotine will be provided throughout the intervention period (24 weeks).
  Interventions: Other: e-cigarette

INTERVENTIONS:
Other: e-cigarette
  Arms: e-cigarette (with 0 mg/ml nicotine); e-cigarette (with 36 mg/ml nicotine); e-cigarette (with 8 mg/ml nicotine)
Other: cigarette substitute
  Arms: cigarette substitute

SUMMARY:
The purpose of this study is to use Randomized Controlled Trial (RCT) methods to examine the influence of novel tobacco products on biomarkers of toxicant exposure and disease risk, reports of adverse events, and concurrent use of other tobacco products. In this case, the novel products are one type of electronic cigarette and an imitation cigarette or cigarette substitute.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65
* Smoke >9 cigarettes per day for at least 1 year
* Smoke regular filtered cigarettes or machine-rolled cigarettes with a filter
* CO measurement >9 ppm at baseline
* No serious quit attempt in the prior 1 month. This includes use of any FDA approved smoking cessation medication (varenicline, bupropion [used specifically as a quitting aid], patch, gum, lozenge, inhaler, and nasal spray) in the past 1 month as an indication of treatment seeking.
* Not planning to quit in the next 6 months
* Interested in reducing cigarette consumption
* Willing to attend visits weekly and monthly over a 9-month period (not planning to move, not planning extended vacation, no planned surgeries)
* Read and write in English
* Able to understand and consent

Exclusion Criteria:

* Pregnant and/or nursing women
* Unstable or significant medical condition in the past 12 months (Recent heart attack or some other heart conditions, stroke, severe angina including high blood pressure if systolic >159 or diastolic >99 observed during screening).
* Immune system disorders, respiratory diseases (exacerbations of asthma or COPD, require oxygen, require oral prednisone), kidney (dialysis) or liver diseases (cirrhosis), or any medical disorder/medication that may affect participant safety or biomarker data.
* Use of any non-cigarette nicotine delivery product (pipe, cigar, dip, chew, snus, hookah, ECIGs, strips, sticks) in the past 7 days
* Uncontrolled mental illness or substance abuse or inpatient treatment for these in the past 6 months
* History of difficulty providing or unwilling to provide blood samples (fainting, poor veins, anxiety)
* No surgery requiring general anesthesia in the past 6 weeks
* Use of an ECIG for 5 or more days in the past 28 days or any use in the past 7 days
* Use of marijuana or any illicit drug/prescription drugs for non-medical use daily/almost daily, or weekly in the past 3 months per NIDA Quick Screen
* Use of hand-rolled, roll your own cigarettes
* Known allergy to propylene glycol or vegetable glycerin
* Other member of household is currently participating/participated in the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
urine carcinogen biomarker of exposure, NNAL | week 24
  changes in NNAL concentration measured at week 0, week 4, week 12, and week 24

SECONDARY OUTCOMES:
urine biomarker of nicotine exposure, cotinine | week 24
  changes in cotinine concentration measured at week 0, week 4, week 12, and week 24
blood, urine, and exhaled breath condensate biomarkers of oxidative stress, glutathione and 8 Isoprostanes | week 24
  changes in oxidative stress biomarker concentrations measured at week 0, week 4, week 12, and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Eissenberg, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Center for the Study of Tobacco Products, Richmond, Virginia

REFERENCES:
- [Derived] Dahal S, Yingst J, Wang X, Cobb CO, Carrillo M, Hrabovsky S, Bascom R, Lopez AA, Kang L, Maloney S, Halquist M, Foulds J, Veldheer S. Changes in cardiovascular disease risk, lung function and other clinical health outcomes when people who smoke use e-cigarettes to reduce cigarette smoking: an exploratory analysis from a randomised placebo-controlled trial. BMJ Open. 2025 Jun 18;15(6):e098005. doi: 10.1136/bmjopen-2024-098005. PMID 40533223
- [Derived] Cobb CO, Budd S, Maldonado G, Imran R, Foulds J, Yingst J, Yen MS, Kang L, Sun S, Hall PB, Chowdhury N, Cohen JE; Randomized Control Trial Methods Workgroup of the Center for the Study of Tobacco Products: Member List. Predictors of attrition in a randomized controlled trial of an electronic nicotine delivery system among people interested in cigarette smoking reduction. Contemp Clin Trials. 2024 Oct;145:107662. doi: 10.1016/j.cct.2024.107662. Epub 2024 Aug 12. PMID 39142511
- [Derived] Cobb CO, Foulds J, Yen MS, Veldheer S, Lopez AA, Yingst JM, Bullen C, Kang L, Eissenberg T; Randomised Control Trial Methods Workgroup of the Center for the Study of Tobacco Products. Effect of an electronic nicotine delivery system with 0, 8, or 36 mg/mL liquid nicotine versus a cigarette substitute on tobacco-related toxicant exposure: a four-arm, parallel-group, randomised, controlled trial. Lancet Respir Med. 2021 Aug;9(8):840-850. doi: 10.1016/S2213-2600(21)00022-9. Epub 2021 Apr 12. PMID 33857436
- [Derived] Lopez AA, Cobb CO, Yingst JM, Veldheer S, Hrabovsky S, Yen MS, Foulds J, Eissenberg T. A transdisciplinary model to inform randomized clinical trial methods for electronic cigarette evaluation. BMC Public Health. 2016 Mar 3;16:217. doi: 10.1186/s12889-016-2792-8. PMID 26941050